CLINICAL TRIAL: NCT00359554
Title: VAXICOL: Effectiveness of Influenza Vaccination of Nursing Home Workers on Mortality of Nursing Home Residents. A Cluster Randomized Trial.
Brief Title: Influenza Vaccination of Nursing Home Workers.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM 05050
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Influenza Disease
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: VAXIGRIPPE

SUMMARY:
The objective of this study is to demonstrate that influenza vaccination of nursing home workers is an effective intervention for reducing mortality of elderly people.

DETAILED DESCRIPTION:
Nursing homes will be randomized within each pair in two arms "incentive to vaccinate", and "do-nothing". In the arm "incentive to vaccinate", vaccination campaigns will be carried out with face-to-face interviews of nursing home workers in order to achieve more than 80% of vaccination coverage. In the "do-nothing", nursing home workers will be vaccinated as usual.

The main endpoint criterion is all-cause mortality of residents. Population sets will be all residents who will be present at start of the influenza season (-2 weeks) or who will be admitted during the influenza season (+ 2 weeks). Onset and end of influenza season will be given by regional influenza surveillance system. Secondary criteria are hospitalizations of residents, morbidity of nursing home workers. A cost-effectiveness ratio of influenza vaccination will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Criteria for nursing home:

* Nursing home whose representative physicians agree to participate, with 50 to 200 residents, located in Paris area, and where the vaccination coverage of nursing home workers was lower than 40% during the previous influenza season (2005).

Criteria for residents:

* All residents who will be present at start of the influenza season (-2 weeks) or who will be admitted during the influenza season (+ 2 weeks).

Exclusion Criteria:

* People before 60 years Not presences in the EHPAD at the time of the beginning of the study (at the moment of the beginning of the epidemic - 2 weeks) or not allowed before the end of the study (before the end of the epidemic + 4, weeks)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2006-09; Study Completion 2007-10

PRIMARY OUTCOMES:
all-cause mortality of residents at one year

SECONDARY OUTCOMES:
hospitalizations of residents,morbidity of nursing home workers.
A cost-effectiveness ratio of influenza vaccination will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice CARRAT, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint Antoine Inserm U707, Paris, France

REFERENCES:
- [Background] Carman WF, Elder AG, Wallace LA, McAulay K, Walker A, Murray GD, Stott DJ. Effects of influenza vaccination of health-care workers on mortality of elderly people in long-term care: a randomised controlled trial. Lancet. 2000 Jan 8;355(9198):93-7. doi: 10.1016/S0140-6736(99)05190-9. PMID 10675165
- [Background] Potter J, Stott DJ, Roberts MA, Elder AG, O'Donnell B, Knight PV, Carman WF. Influenza vaccination of health care workers in long-term-care hospitals reduces the mortality of elderly patients. J Infect Dis. 1997 Jan;175(1):1-6. doi: 10.1093/infdis/175.1.1. PMID 8985189
- [Background] Thomas RE, Jefferson TO, Demicheli V, Rivetti D. Influenza vaccination for health-care workers who work with elderly people in institutions: a systematic review. Lancet Infect Dis. 2006 May;6(5):273-9. doi: 10.1016/S1473-3099(06)70462-5. PMID 16631547